CLINICAL TRIAL: NCT03887650
Title: LIBERATE - LIposomal Bupivacaine vERsus Adjuncts in Total shouldErs: A Randomized Controlled Trial of Injection at the Brachial Plexus
Brief Title: LIBERATE - LIposomal Bupivacaine vERsus Adjuncts in Total shouldErs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Kevin Finkel, Principal Investigator, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HHC-2018-0231
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Post-operative Pain; Total Shoulder Arthroplasty; Osteoarthritis of the Shoulder; Pain Management
Keywords: Brachial Plexus; Liposomal Bupivacaine; Dexamethasone; Interscalene; Bupivacaine; Shoulder Arthroplasty; Regional anesthesia; Exparel
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Epinephrine

STUDY DESIGN:
Intervention Model Description: single-center, prospective, randomized controlled cross-sectional study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal Bupivacaine 1.3% (Experimental): 10mL Liposomal Bupivacaine 1.3% (133 mg) mixed with 10mL of 0.5% Bupivacaine (total volume 20mL) in single injection interscalene brachial plexus block
  Interventions: Drug: Liposomal Bupivicaine 1.3%
- Bupivacaine 0.5% with Adjuncts (Active Comparator): 20mL 0.5% Bupivacaine with 5 mg PF dexamethasone and 5 mcg epinephrine (total volume 20.5mL) in single injection interscalene brachial plexus block
  Interventions: Drug: Bupivacaine 0.5%

INTERVENTIONS:
Drug: Liposomal Bupivicaine 1.3% — 10mL Liposomal Bupivacaine 1.3% (133 mg) mixed with 10mL of 0.5% Bupivacaine (total volume 20mL) in single injection interscalene brachial plexus block
  Arms: Liposomal Bupivacaine 1.3%
Drug: Bupivacaine 0.5% — 20mL 0.5% Bupivacaine with 5 mg PF dexamethasone and 5 mcg epinephrine (total volume 20.5mL) in single injection interscalene brachial plexus block
  Other Names: epinephrine; dexamethasone preservative-free
  Arms: Bupivacaine 0.5% with Adjuncts

SUMMARY:
This will be a single-center, prospective, randomized controlled cross-sectional study comparing interscalene brachial plexus block with liposomal bupivacaine versus bupivacaine with epinephrine and PF dexamethasone in patients undergoing primary shoulder arthroplasty. Primary endpoint will be total opioid consumption in the first three post-operative days.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18 years;
* Lack of language barrier;
* Informed consent obtained;
* Presenting for primary total shoulder arthroplasty (TSA), both anatomic and reverse, by a specialty-trained surgeon;
* American Society of Anesthesiology (ASA) physical status score I- III

Exclusion Criteria:

* Presence of a language barrier;
* Inability to complete telephone and/or paper questionnaire;
* Lack of consent;
* Allergy to local anesthetic;
* Chronic pain syndrome and/or preoperative opioid use > 50 MME per day (including extended-release formulations and methadone);
* Preoperative consultation to chronic pain service;
* History of (<3 months) or current substance abuse, including any illicit drugs or excessive alcohol consumption as defined by the Office of Disease Prevention and Health Promotion (4 or more drinks per day or 8 or more drinks per week for women and 5 or more drinks per day or 15 or more drinks per week for men);
* Baseline peripheral neuropathy of the brachial plexus;
* Contraindication to receiving single shot peripheral nerve blockade; including antithrombotic medications as per most recent American Society of Regional - - -Anesthesiology (ASRA) guidelines 17 , coagulopathy or coagulation disorder, or infection at injection site;
* Severe chronic obstructive pulmonary disease (COPD) or other significant pulmonary disease where interscalene nerve block would be contraindicated due to concern for respiratory failure from phrenic nerve palsy;
* Weight < 45 kg, given concern for local anesthetic toxicity at dosages given for the study; ASA score IV-V;
* Revision arthroplasty;
* Anatomic abnormality that limits or prevents the patient from receiving an interscalene nerve block;
* Pregnant, nursing, or planning to become pregnant during the study or within 1 month after the shoulder replacement surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Finkel, MD, Principal Investigator — Hartford Hospital
Locations (1):
- The Bone and Joint Institute at Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Vieira PA, Pulai I, Tsao GC, Manikantan P, Keller B, Connelly NR. Dexamethasone with bupivacaine increases duration of analgesia in ultrasound-guided interscalene brachial plexus blockade. Eur J Anaesthesiol. 2010 Mar;27(3):285-8. doi: 10.1097/EJA.0b013e3283350c38. PMID 20009936
- [Background] Movafegh A, Razazian M, Hajimaohamadi F, Meysamie A. Dexamethasone added to lidocaine prolongs axillary brachial plexus blockade. Anesth Analg. 2006 Jan;102(1):263-7. doi: 10.1213/01.ane.0000189055.06729.0a. PMID 16368840
- [Background] Parrington SJ, O'Donnell D, Chan VW, Brown-Shreves D, Subramanyam R, Qu M, Brull R. Dexamethasone added to mepivacaine prolongs the duration of analgesia after supraclavicular brachial plexus blockade. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):422-6. doi: 10.1097/AAP.0b013e3181e85eb9. PMID 20814282
- [Background] Rasmussen SB, Saied NN, Bowens C Jr, Mercaldo ND, Schildcrout JS, Malchow RJ. Duration of upper and lower extremity peripheral nerve blockade is prolonged with dexamethasone when added to ropivacaine: a retrospective database analysis. Pain Med. 2013 Aug;14(8):1239-47. doi: 10.1111/pme.12150. Epub 2013 Jun 11. PMID 23755801
- [Background] McLaughlin DC, Cheah JW, Aleshi P, Zhang AL, Ma CB, Feeley BT. Multimodal analgesia decreases opioid consumption after shoulder arthroplasty: a prospective cohort study. J Shoulder Elbow Surg. 2018 Apr;27(4):686-691. doi: 10.1016/j.jse.2017.11.015. Epub 2018 Jan 3. PMID 29305103
- [Background] Candiotti K. Liposomal bupivacaine: an innovative nonopioid local analgesic for the management of postsurgical pain. Pharmacotherapy. 2012 Sep;32(9 Suppl):19S-26S. doi: 10.1002/j.1875-9114.2012.01183.x. PMID 22956491
- [Background] Abildgaard JT, Lonergan KT, Tolan SJ, Kissenberth MJ, Hawkins RJ, Washburn R 3rd, Adams KJ, Long CD, Shealy EC, Motley JR, Tokish JM. Liposomal bupivacaine versus indwelling interscalene nerve block for postoperative pain control in shoulder arthroplasty: a prospective randomized controlled trial. J Shoulder Elbow Surg. 2017 Jul;26(7):1175-1181. doi: 10.1016/j.jse.2017.03.012. Epub 2017 May 4. PMID 28479257
- [Background] Hannan CV, Albrecht MJ, Petersen SA, Srikumaran U. Liposomal Bupivacaine vs Interscalene Nerve Block for Pain Control After Shoulder Arthroplasty: A Retrospective Cohort Analysis. Am J Orthop (Belle Mead NJ). 2016 Nov/Dec;45(7):424-430. PMID 28005096
- [Background] Wang K, Zhang HX. Liposomal bupivacaine versus interscalene nerve block for pain control after total shoulder arthroplasty: A systematic review and meta-analysis. Int J Surg. 2017 Oct;46:61-70. doi: 10.1016/j.ijsu.2017.08.569. Epub 2017 Aug 24. PMID 28843463
- [Background] Schroer WC, Diesfeld PG, LeMarr AR, Morton DJ, Reedy ME. Does Extended-Release Liposomal Bupivacaine Better Control Pain Than Bupivacaine After Total Knee Arthroplasty (TKA)? A Prospective, Randomized Clinical Trial. J Arthroplasty. 2015 Sep;30(9 Suppl):64-7. doi: 10.1016/j.arth.2015.01.059. Epub 2015 Jun 3. PMID 26117072
- [Background] Vandepitte C, Kuroda M, Witvrouw R, Anne L, Bellemans J, Corten K, Vanelderen P, Mesotten D, Leunen I, Heylen M, Van Boxstael S, Golebiewski M, Van de Velde M, Knezevic NN, Hadzic A. Addition of Liposome Bupivacaine to Bupivacaine HCl Versus Bupivacaine HCl Alone for Interscalene Brachial Plexus Block in Patients Having Major Shoulder Surgery. Reg Anesth Pain Med. 2017 May/Jun;42(3):334-341. doi: 10.1097/AAP.0000000000000560. PMID 28157791

RESULTS

PARTICIPANT FLOW:
Period: Preoperative-48 Hours Postoperative
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts
Started | 45 | 45
Completed | 45 | 44
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: 48-96 Hours Postoperative
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts
Started | 45 (A patient who was lost to follow-up from the previous period came back for this period of the study) | 44
Completed | 45 | 42
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: 60 Postoperative Days
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts
Started | 45 | 42
Completed | 44 | 42
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72 [66.5 to 77.0] | 73 [66.5 to 78.0] | 73 [66.75 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 23 | 22 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 44 | 44 | 88
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 44 | 42 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 31.30 [27.25 to 33.65] | 31.60 [27.00 to 35.850] | 31.35 [27.25 to 34.23]
ASA Physical Status Classification [Median (Inter-Quartile Range); unit: units on a scale] — American Society of Anesthesiologists (ASA) physical status classification. ASA scale ranges (1-6), where 1 is the best while 6 is the worst ASA I = A normal healthy patient ASA II = A patient with mild systemic disease ASA III = A patient with severe systemic disease ASA IV = A patient with severe systemic disease that is a constant threat to life ASA V = A moribund patient who is not expected to survive without the operation ASA VI = A declared brain-dead patient whose organs are being removed for donor purposes
  units on a scale | 2 [2 to 3] | 2 [2 to 3] | 2 [2 to 3]
Preoperative shoulder pain [Count of Participants; unit: Participants]
  None | 12 | 11 | 23
  Mild | 16 | 20 | 36
  Moderate | 15 | 7 | 22
  Severe | 2 | 7 | 9
Comorbidities [Count of Participants; unit: Participants]
  Diabetes Miletus : yes | 6 | 9 | 15
  Diabetes Miletus : no | 39 | 36 | 75
  Hyperlipidemia : yes | 26 | 25 | 51
  Hyperlipidemia : no | 19 | 20 | 39
  Hypertension : yes | 29 | 25 | 54
  Hypertension : no | 16 | 20 | 36
  COPD : yes | 0 | 2 | 2
  COPD : no | 45 | 43 | 88
  RA : yes | 0 | 3 | 3
  RA : no | 45 | 42 | 87
  Opioids at home : yes | 3 | 6 | 9
  Opioids at home : no | 42 | 39 | 81

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Consumption
Description: Total opioids used for the first 120 postoperative hours after TSA, standardized to morphine milligram equivalents (MMEs)
Time Frame: Up to 120 postoperative hours
Population: 3 patients withdrew from Bupivacaine 0.5% with Adjuncts group.
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts
Number analyzed (Participants) | 45 | 42
MME | 71.25 [43.00 to 120.00] | 90.30 [57.37 to 133.43]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = 0.127, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Time to First Opioid Medication
Description: From block time to the first dose of opioids given, measured in hours.
Time Frame: from the time of the block injection until discharge, assessed up to 72 postoperative hours.
Population: Missing data for 2 patients from the Liposomal Bupivacaine 1.3% group. 3 patients withdrew consents from the Bupivacaine 0.5% with Adjuncts group.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts
Number analyzed (Participants) | 43 | 42
hours | 10.5667 [5.800 to 20.850] | 12.025 [4.404 to 21.983]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .975, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Pain Assessment at Post Anesthesia Care Unit (PACU)-96 Postoperative Hours
Description: Pain assessment is categorized as minimum, maximum, and average pain scores reported by patients using questions from the Modified Brief Pain Inventory-short form (MBPI-SF) during the following intervals; PACU-24, 24-48, 48-72, and 72-96 postoperative hours, and at day 60. This form collected minimum, maximum, and average on a numeric pain scale (0-10) where 0 is no pain and 10 is the worst pain.
Time Frame: 24, 24-48, 48-72, and 72-96 hours postoperation, and at day 60
Population: Three patients withdrew consent from the control group (Bupivacaine 0.5% with adjuncts) and one from the liposomal bupivacaine group. The rest is missing data from lost to follow-up.
Measure: Median (Inter-Quartile Range); unit: units on a scale 0-10
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts
Number analyzed (Participants) | 45 | 45
units on a scale 0-10
  PACU | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 1.50]
  PACU-24 hours Minimum | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 0.00]
  PACU-24 hours Maximum | 2.00 [0.00 to 4.50] | 1.00 [0.00 to 4.50]
  PACU-24 hours Average | 1.00 [0.00 to 2.00] | 0.00 [0.00 to 3.50]
  24-48 hours Minimum: number analyzed (Participants) | 44 | 44
  24-48 hours Minimum | 0.00 [0.00 to 2.00] | 2.00 [0.00 to 3.75]
  24-48 hours Maximum: number analyzed (Participants) | 44 | 44
  24-48 hours Maximum | 4.50 [1.00 to 6.00] | 7.00 [5.00 to 8.00]
  24-48 hours Average: number analyzed (Participants) | 44 | 44
  24-48 hours Average | 2.00 [0.00 to 3.75] | 4.00 [3.00 to 5.00]
  48-72 hours Minimum: number analyzed (Participants) | 41 | 41
  48-72 hours Minimum | 1.00 [0.00 to 2.00] | 2.00 [1.00 to 3.00]
  48-72 hours Maximum: number analyzed (Participants) | 41 | 41
  48-72 hours Maximum | 4.00 [1.75 to 6.00] | 6.00 [4.50 to 7.00]
  48-72 hours Average: number analyzed (Participants) | 41 | 41
  48-72 hours Average | 2.00 [1.00 to 3.25] | 3.00 [2.00 to 5.00]
  72-96 hours Minimum: number analyzed (Participants) | 41 | 41
  72-96 hours Minimum | 0.50 [0.00 to 2.00] | 2.00 [0.00 to 2.00]
  72-96 hours Maximum: number analyzed (Participants) | 41 | 41
  72-96 hours Maximum | 4.00 [1.75 to 5.25] | 5.00 [4.00 to 7.0]
  72-96 hours Average: number analyzed (Participants) | 41 | 41
  72-96 hours Average | 2.00 [1.00 to 3.00] | 3.00 [2.00 to 4.00]
  60 days postoperative Maximum: number analyzed (Participants) | 40 | 40
  60 days postoperative Maximum | 5.00 [2.00 to 6.00] | 6.00 [4.25 to 8.00]
  60 days postoperative Average: number analyzed (Participants) | 40 | 40
  60 days postoperative Average | 1.00 [0.25 to 3.00] | 2.00 [1.00 to 3.00]
  60 days postoperative Minimum: number analyzed (Participants) | 40 | 40
  60 days postoperative Minimum | 0.00 [0.00 to 0.75] | 0.00 [0.00 to 1.00]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .852, Wilcoxon (Mann-Whitney) — PACU pain scores
Statistical Analysis 2: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .661, Wilcoxon (Mann-Whitney) — For (PACU-24) minimum pain scores
Statistical Analysis 3: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .747, Wilcoxon (Mann-Whitney) — For (PACU-24 hr.) maximum pain score
Statistical Analysis 4: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .604, Wilcoxon (Mann-Whitney) — For (PACU-24 hr) average pain scores
Statistical Analysis 5: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .002, Wilcoxon (Mann-Whitney) — (24-48 hr) minimum pain scores
Statistical Analysis 6: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney) — For (24-48 hr) maximum pain scores
Statistical Analysis 7: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney) — For (24-48 hr) average pain scores
Statistical Analysis 8: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .011, Wilcoxon (Mann-Whitney) — (48-72 hr) minimum pain scores
Statistical Analysis 9: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .001, Wilcoxon (Mann-Whitney) — (48-72 hr) maximum pain scores
Statistical Analysis 10: Comparison: Liposomal Bupivacaine 1.3%; Test type: Superiority; p = .003, Wilcoxon (Mann-Whitney) — (48-72 hr) average pain scores
Statistical Analysis 11: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .230, Wilcoxon (Mann-Whitney) — For (72-96 hr) minimum pain scores
Statistical Analysis 12: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .007, Wilcoxon (Mann-Whitney) — For (72-96 hr) maximum pain scores
Statistical Analysis 13: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .011, Wilcoxon (Mann-Whitney) — For (72-96 hr) average pain scores
Statistical Analysis 14: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .378, Wilcoxon (Mann-Whitney) — For (postoperative day 60) minimum pain scores
Statistical Analysis 15: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .001, Wilcoxon (Mann-Whitney) — For (postoperative day 60) maximum pain scores
Statistical Analysis 16: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .403, Wilcoxon (Mann-Whitney) — For (postoperative day 60) average pain scores

4. Secondary Outcome: Hospital Length-of-stay
Description: From the date and time of admission to the date and time of discharge, Measured in hours.
Time Frame: From the date of admission until discharge, assessed up to 72 hours.
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts
Number analyzed (Participants) | 45 | 45
hour | 31.05 [29.67 to 32.53] | 31.63 [30.63 to 36.58]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .112, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Assessment of Patient Overall Satisfaction With Pain Control
Description: Patient overall satisfaction with pain control was assessed two times; on the fourth and the 60th postoperative days. It was assessed using a numeric scale (0-10) where 0 is very dissatisfied while 10 is extremely satisfied. The results indicated only the percentage of participants who reported a 10/10 satisfaction rate.
Time Frame: POD4 - 60 days
Population: One patient withdrew consent from the Liposomal group just prior to 60 postoperative days, and three patients withdrew consent from the control group at the end of days 2, 3, and 4. The other missing data is from patients who lost to follow up from both groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts
Number analyzed (Participants) | 45 | 42
Participants
  POD4: 10/10 | 32 | 24
  POD4: below 10 | 9 | 17
  POD4: Missing data | 4 | 1
  POD60: number analyzed (Participants) | 44 | 42
  POD60: 10/10 | 27 | 28
  POD60: below 10 | 12 | 13
  POD60: Missing data | 5 | 1
Statistical Analysis 1: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = 0.096, Fisher Exact — P-Value for POD4; Fisher's Exact for POD4
Statistical Analysis 2: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = 1.0, Chi-squared — For POD60; Chi-squared for POD60

6. Secondary Outcome: Incidence of Distress From Block Numbness
Description: On a distress scale of (0 -10) with 0 = not at all and 10 = very much distressed, the scores were gathered and the results are grouped to show the percentage of either the presence of distress (any positive score) or no distress, assessed at two times; at the PACU and the second postoperative day.
Time Frame: At PACU and Postoperative day 2
Population: Although one patient from the control group decided to withdraw consent at the end of the second day following surgery, their data was included for this outcome as the withdrawal happened after collection. However, there was some missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts
Number analyzed (Participants) | 45 | 45
Participants
  PACU distress: No distress | 31 | 31
  PACU distress: any distress | 14 | 14
  PACU distress: Missing data | 0 | 0
  POD2 Distress: No distress | 32 | 31
  POD2 Distress: any distress | 12 | 12
  POD2 Distress: Missing data | 1 | 2
Statistical Analysis 1: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = 1.0, Chi-squared — Any distress on PACU
Statistical Analysis 2: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .947, Chi-squared — Postoperative day 2

7. Secondary Outcome: Duration of Sensory Nerve Block
Description: Using the sensory assessment test, the results show the percentage of participants who had the return of first sensation and full sensation either on Day 1, after Day 1 (day 2 to 60), and at postoperative day 60.
Time Frame: Day 1, after Day 1 (day 2 to 60), and at postoperative day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts
Number analyzed (Participants) | 45 | 45
Participants
  Full sensation: Returned on day 1 after the block | 11 | 11
  Full sensation: Returned on day 2-60 | 27 | 27
  Full sensation: Not by day 60 | 0 | 2
  Full sensation: Missing data | 7 | 5
  First sensation: Returned on day 1 after the block | 35 | 33
  First sensation: Returned on day 2-60 | 9 | 10
  First sensation: Not by day 60 | 0 | 0
  First sensation: Missing data | 1 | 2
Statistical Analysis 1: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .441, Fishers Freeman Halton — Full sensation
Statistical Analysis 2: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .691, Fishers Freeman Halton — First sensation

8. Secondary Outcome: Day of the Final Opioids Used
Description: The postoperative day that patients in each group took their last opioid, from the end of surgery up to 96 postoperative hours.
Time Frame: 0-96 postoperative hours
Population: Three patients were missing from (Bupivacaine 0.5% with Adjuncts) group because of withdrawal.
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts
Number analyzed (Participants) | 45 | 42
day | 4 [1.5 to 4] | 4 [1 to 4]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .876, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Motor Recovery
Description: The Motor function was assessed by shoulder abduction and elbow flexion using the Oxford scale of muscle strength grading (Muscle Grading Scores 0-5):
  0= No detectable muscle contraction (visible or palpation)
  1. Detectable contraction (visible or palpation), but no movement achieved
  2. Limb movement achieved, but unable to move against gravity
  3. Limb movement against the resistance of gravity
  4. Limb movement against gravity and external resistance
  5. Normal strength
  The results were grouped to show the return of any movement at the PACU, Day 1, after Day 1 (day2-60), and on day 60. And the return of full movement between day 2 and 60 and at day 60, in addition to the missing data.
Time Frame: PACU, Day 1, after Day 1 (day 2 and 60), and at postoperative day 60.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts
Number analyzed (Participants) | 45 | 45
Participants
  Any movement in PACU | 1 | 11
  Any movement in day1 | 4 | 3
  Any movement after day1 | 38 | 29
  Any movement missing data | 2 | 2
  Return of full movement day 2-60 | 32 | 31
  Not yet by day 60 | 3 | 6
  Return of full movement missing data | 10 | 8
Statistical Analysis 1: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .011, Fisher' Freeman Halton — Any movement
Statistical Analysis 2: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .536, Fishers Freeman Halton — Full movement

10. Other Pre Specified Outcome: Total Amount of Opioid Consumed During the Indicated Time Periods
Description: Opioid use was calculated using the Morphine MilliEquevalent per day, this was assessed daily during the postoperative period, 0-24, 24-48, 48-72, and 72-120 postoperative hours.
Time Frame: 0-24, 24-48, 48-72, and 72-120 postoperative hours.
Population: One patient withdrew consent on the second postoperative day from the control group, then two patients withdrew on the third and fourth postoperative days from the control group.
Measure: Median (Inter-Quartile Range); unit: MME/day
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts
Number analyzed (Participants) | 45 | 45
MME/day
  0-24 hours | 25.00 [25.00 to 39.37] | 25.00 [25.00 to 37.50]
  24-48 hours | 16.00 [0.00 to 38.75] | 23.25 [9.75 to 39.37]
  48-72 hours: number analyzed (Participants) | 45 | 44
  48-72 hours | 2.00 [0.00 to 8.00] | 5.00 [0.00 to 15.00]
  72-120 hours: number analyzed (Participants) | 44 | 42
  72-120 hours | 10.00 [0.00 to 27.00] | 15.00 [0.00 to 37.50]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .648, Wilcoxon (Mann-Whitney) — MME 0-24
Statistical Analysis 2: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .285, Wilcoxon (Mann-Whitney) — MME24-48
Statistical Analysis 3: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .122, Wilcoxon (Mann-Whitney) — MME48-72
Statistical Analysis 4: Comparison: Liposomal Bupivacaine 1.3% vs Bupivacaine 0.5% With Adjuncts; Test type: Superiority; p = .367, Wilcoxon (Mann-Whitney) — MME 72-120

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 60 postoperative days.
Arm/Group | Liposomal Bupivacaine 1.3% | Bupivacaine 0.5% With Adjuncts
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 18/45 | 21/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Bupivacaine 1.3% (N=45) | Bupivacaine 0.5% With Adjuncts (N=45)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Rash around the block site
Swelling (Surgical and medical procedures) | 1 (1) | 0 (0) — Swelling of shoulder surgical site
Inflammation (Surgical and medical procedures) | 1 (1) | 0 (0)
Bruising (Surgical and medical procedures) | 5 (5) | 3 (3)
Ringing in ears (Ear and labyrinth disorders) | 1 (1) | 1 (1) — On the block side
Numbness and tingling (Nervous system disorders) | 1 (1) | 0 (0) — Of same surgery side shoulder and arm
Nausea and vomiting (General disorders) | 8 (8) | 16 (16)

LIMITATIONS AND CAVEATS:
Opioid consumption was subjected to patient recall and reporting bias. Patients were advised by surgery clinics to limit opioid intake postoperatively, which might indirectly limit opioid use and made it more difficult to show a difference. The study was double-blinded, the anesthesiologists who performed the block, were unblinded due to the difference in the physical appearance of the study drugs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT03887650/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT03887650/ICF_001.pdf